CLINICAL TRIAL: NCT00144326
Title: A Randomised, Double-blind, Placebo-controlled, 12 Week Trial to Evaluate the Effect, of Tiotropium Inhalation Capsules on the Magnitude of Exercise, Measured Using an Accelerometer, in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Randomised, Double-blind, Placebo-controlled, 12 Week Trial to Evaluate the Effect of Tiotropium Inhalation Capsules (Spiriva) on the Magnitude of Exercise, Measured Using an Accelerometer, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.269
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium Bromide
Drug: Placebo

SUMMARY:
The objective of this study is to determine if tiotropium (Spiriva, Bromuro de Tiotropio) 18 mcg once daily by oral inhalation compared to placebo increases the magnitude of daily physical activity observed in COPD patients, measured using an accelerometer.

DETAILED DESCRIPTION:
This is a 3 month, multicentre, randomised, double-blind, placebo controlled, parallel group study to compare with placebo the long-term effect of tiotropium inhalation capsules on daily physical activity in patients with COPD.

The drugs will be administered in the form of inhalation capsules of tiotropium or placebo, taken once daily in the morning.

The record of daily physical activity using the accelerometer will be carried out at all study visits other than Visit 1. The accelerometer will be used for the five day period, from Thursday to Monday, closest to the corresponding visit.

The pulmonary function tests will be carried out at Visit 1 (screening visit), Visit 2 (baseline visit) and study visits (Visits 3 to 5) with the restrictions detailed at the trial protocol.

Study Hypothesis:

The null hypothesis is that there is no difference between tiotropium (Spiriva) and placebo regarding the magnitude of exercise measured with an accelerometer. The alternative hypothesis is that there is a difference between tiotropium (Spiriva) and placebo regarding the magnitude of exercise measured with an accelerometer.

Comparison(s):

The difference in physical activity measured in vector magnitude units (VMUs) by the triaxial Stayhealthy RT3 accelerometer at the end of the three month treatment period compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* All patients must sign an Informed Consent Form consistent with ICH-GPC guidelines prior to participation in the trial
* Diagnosis of COPD and meets the following spirometric criteria:

  * The patients must present with relatively stable* airway obstruction
  * An FEV1 <= 65% of the predicted normal value and an FEV1 <= 70% of the FVC, at visit 1 (screening). This must be confirmed at visit 2 (baseline).
* Male or female patients of 40 years of age or older.
* The patients must be smokers or ex-smokers with a history of having smoked at least 10 pack-years.
* The patients must be able to carry out all the tests related to the study, including the slow and forced spirometry and the 6 minute walk test, exactly as required in the protocol.
* The patients must be able to inhale the medication by means of the HandiHaler.

Exclusion Criteria:

* Those patients with significant diseases other than COPD will be excluded.
* Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during the study.
* Patients with any respiratory tract infection in the past six weeks prior to the screening visit (Visit 1) or during the run-in period, prior to Visit 2 (baseline).
* Patients with a past history of asthma, allergic rhinitis or atopy, or who present a total eosinophil count >= 600 mm3. No new eosinophil count will be undertaken in these patients.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10

PRIMARY OUTCOMES:
Primary endpoint: The primary efficacy variable will be the difference in physical activity measured in vector magnitude units (VMUs) by the triaxial Stayhealthy RT3 accelerometer at the end of the three month treatment period compared to placebo.

SECONDARY OUTCOMES:
Pulmonary function tests, distance covered in the 6MWD, Modified Borg Dyspnea scale, QoL measured by the CRQ, use of rescue salbutamol, and safety variables.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Spain S.A.
Locations (26):
- Canada (6):
  - 1796 Summer Street, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Respiratory/ Research Lab, Toronto, Ontario
  - Montreal Chest Institute of the Royal Victoria Hospital, Montreal, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Department of Respiratory Medicine, Saskatoon, Saskatchewan
- Germany (9):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Klinik III für Innere Medizin/ Pneumologie, Cologne
  - Krankenhaus Donaustauf, Donaustauf
  - Boehringer Ingelheim Investigational Site, Fürth
  - Inamed Research GmbH & Co. KG, Gauting
  - Pneumologisches Forschungsinstitut GmbH, Großhansdorf
  - Pneumologisches Forschungsinstitut GmbH am Krankenhaus, Hamburg
  - Allergomedic, Hanover
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
- Spain (11):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares (Madrid)
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Centro de Asistencia Primaria de Campdevanol, Campdevànol (Girona)
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reína Sofía, Córdoba
  - Hospital General de Elche, Elche (Alicante)
  - Hospital Ntra. Sra. de Meritxell, Escaldes-Engordany
  - Centro de Asistencia Primaria de la Roca, La Roca Del Vallés (Barcelona)
  - Hospital de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Vírgen de la Victoria, Málaga